CLINICAL TRIAL: NCT03158753
Title: Perfusion Index and Pain in Ankle Surgery - an Exploratory Study
Brief Title: Perfusion Index and Pain in Ankle Surgery
Acronym: PIPA
Status: Completed | Type: Observational
Sponsor: Rune Sort (Other)
Responsible Party: Sponsor-Investigator, Rune Sort, Principal Investigator, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: PIPA study
Record Dates: First submitted 2017-05-03; First posted 2017-05-18 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Pain, Postoperative; Ankle Fractures
MeSH Terms: conditions — Pain, Postoperative; Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perfusion index (PI) measured via a pulse oximeter has been shown to correlate with activation of the sympathetic nervous system, such as by pain stimulation, as a result of involuntary contraction of the arterioles. Thus PI holds potential for use as a tool for "objective pain measurement", although its practical usefulness and dependability as such have not previously been investigated.

The investigators aim to explore associations between changes in PI and onset of pain following cessation of regional anaesthesia in alert patients following ankle fracture surgery.

Methods:

The investigators report an exploratory, observational analysis of prospectively gathered PI data from patients undergoing regional anaesthesia with spinal or peripheral nerve block for ankle fracture surgery as participants of the randomised AnAnkle Trial (EudraCT: 2015-001108-76). PI is measured on an unaffected extremity in approximately 20 consecutive patients already included in the AnAnkle Trial at Herlev University Hospital, evenly distributed between spinal anaesthesia (SA) and peripheral nerve block (PNB).

Both anaesthesia forms and pain medication regimes are standardised as part of AnAnkle Trial and participants register pain scores on a 0-10 numeric rating scale every three hours and register the time of cessation of anaesthesia identified by return of sensation to the ankle. Morphine consumption is also registered.

The investigators will explore correlations of changes in PI to increases in pain upon cessation of the regional anaesthesia and, secondly, differences in cessation related PI changes with SA versus PNB.

Ethics:

All participants have already given informed, written consent for use of this data for the AnAnkle Trial. All necessary ethical and legislative approvals have been obtained for initiation of AnAnkle Trial in July 2015.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for internal fixation of an ankle fracture
* Age > 18 years
* Ability to read and understand Danish and give informed written consent

Exclusion Criteria:

* Allergy towards NSAID, paracetamol, morphine or local anaesthetics
* Bodyweight < 52 kg; to avoid toxic doses of local anaesthetics
* Contraindications for SA
* Current gastro-intestinal bleeding
* Proximal fibular fracture or multitrauma / other simultaneous fractures
* Cognitive or psychiatric dysfunction or alcohol/narcotic substance abuse causing expected inability to comply with study protocol
* No available anaesthesiologist with PNB capability at scheduled time of operation
* Neuropathy / neurological dysfunction in the lower extremities
* Habitual daily use of opioids
* Pregnancy or breastfeeding
* Infection at anaesthesia injection site
* Nephropathy requiring dialysis
* Acute porphyria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the AnAnkle Trial at Herlev University Hospital.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
PI changes with rebound pain | 1 hour prior to 6 hours post cessation of regional anaesthesia effect
  Correlation of changes in PI to pain upon cessation of the regional anaesthesia

SECONDARY OUTCOMES:
PI changes in relation to anaesthesia modality | 1 hour prior to 6 hours post cessation of regional anaesthesia effect
  Differences in cessation related PI changes between spinal anaesthesia and PNBs
Timing of PI changes | 1 hour prior to 6 hours post cessation of regional anaesthesia effect
  Exploration of timing of the PI changes related to patient reported cessation of regional anaesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Herlev, Denmark